CLINICAL TRIAL: NCT01598012
Title: The Efficacy of Ayurved Siriraj Prasaplai for Treatment Primary Dysmenorrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R015535011; (IO)R015535011 (Other Grant/Funding Number: Siriraj Research Development Fund)
Record Dates: First submitted 2012-04-09; First posted 2012-05-15 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Primary Dysmenorrhea
Keywords: Ayurved Siriraj Prasaplai; primary dysmenorrhea
MeSH Terms: interventions — Mefenamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ayurved Siriraj Prasaplai (Experimental)
  Interventions: Drug: Ayurved Siriraj Prasaplai with or without mefenamic acid
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo with or without mefenamic acid

INTERVENTIONS:
Drug: Ayurved Siriraj Prasaplai with or without mefenamic acid — Prasaplai in capsule, 2 cap three times a day for 3 days. Mefenamic acid 500 mg prn for severe pain (as rescue medication)
  Other Names: Ponstan
  Arms: Ayurved Siriraj Prasaplai
Drug: Placebo with or without mefenamic acid — Placebo in capsule (physically identical appearance as Prasaplai) 2 cap three times a day for 3 days. Mefenamic acid 500 mg prn for severe pain, every 6 hours (rescue medication)
  Other Names: Ponstan
  Arms: placebo

SUMMARY:
Ayurved Siriraj Prasaplai is a Thai traditional herbal drug for pain treatment. Mostly it was used for antipain during menstruation or dysmenorrhea. This drug has been described by alternative medical doctor for treatment of primary dysmenorrhea for more than 10 years and showed clinical satisfied response. From review about this agent, it does not have clinical trial to prove its efficacy. So the author produce this research to study in efficacy of Ayurved Siriraj Prasaplai.

DETAILED DESCRIPTION:
The participants were allocated in the study by block randomization and double blind. In experiment-group was treated with Ayurved Siriraj Prasaplai and control-group was treated with placebo (non-active agent). Both of drug was made in the same appearance of capsule (size and color). The participants have to start the drug when they have menstruation after that the dosage is 2 capsules for 3 times per day (after-meal) continue to 3 days. The participant have to record pain score (minimal/maximal/mean score) and multidimensional score in daily card, side effect and satisfaction. If the participant couldn't tolerate the pain, they could break the pain with mefenamic acid. They have record number of mefenamic acid which they used too. This study evaluate in only one cycle. After complete record, the participant come back to investigator for sending the report.

ELIGIBILITY:
Inclusion Criteria:

* Woman who is diagnosed of primary dysmenorrhea.
* Woman who has regular menstruation.
* woman who has numeric rating score for pain during menstruation (dysmenorrhea) more than score 5 and continuous for 3 menstrual cycle.
* Woman who want to participate in this study.

Exclusion Criteria:

* Woman who has allergic history for herbal or other components in Ayurved Siriraj Prasaplai drug.
* Woman who has hormonal contraception.
* Woman who has other diseases which is caused of abdominal pain.
* Breast feeding woman

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pain score between experimental and placebo group | 1 year
  Compare pain score by using numeric rating scale (NRS) between the group of women who recieve Ayurved Siriraj Prasaplai with placebo group.

SECONDARY OUTCOMES:
To study about adverse effects of Ayurved Siriraj Prasaplai | 1 year
  To study about adverse effects such as skin rash, nausea vomitting, palpitation, jaundice, hypersensitivity symptoms during treatment with Ayurved Siriraj Prasaplai or placebo.
Number of mefenamic acid for breaking pain during study of both group | 1 year
  During experiment if participant couldn't tolerate the pain which be treated with Ayurved Siriraj Prasaplai or placebo, they could have breaking pain(rescue treatment) with mefenamic acid. Then the participant have to record the number of mefenamic acid and timing which they used in record form.

CONTACTS AND LOCATIONS:
Overall Officials: Thanyarat Wongwananuruk, MD., Principal Investigator — Gynecologic Endocrinology Unit, Department of Obstetric and Gynecology
Locations (1):
- Gynecologic Endocrinology Unit, Department of Obstetric and Gynecology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- See also: Siriraj Institutional Review board (SIRB) — http://www.si.mahidol.ac.th/Th/division/sirb/